CLINICAL TRIAL: NCT00859196
Title: A Randomized, Double-blind, Single Centre, Placebo-controlled Pilot Study to Assess on a Molecular Level the Influence of a 5 % Dexpanthenol Ointment in Subjects With Previously Injured Skin by Investigation of Skin Biopsies
Brief Title: Study to Assess on a Molecular Level the Influence of a 5 % Dexpanthenol Ointment in Subjects With Superficial Injuries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 13069; 2008-002069-30 (EudraCT Number)
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Wound Healing; Cell Proliferation; Gene Expression
Keywords: Wound healing; Cell proliferation; Gene expression
MeSH Terms: conditions — Hyperplasia | interventions — dexpanthenol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Dexpanthenol (BAY81-2996)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexpanthenol (BAY81-2996) — Test product and the respective placebo will be applied to previously wounded test areas and the surrounding skin (approx. 3 cm2). After a certain time the second skin biopsy will be taken from the treated test areas. The skin biopsies will be analysed via micro array.
  Arms: Arm 1
Drug: Placebo — Test product and the respective placebo will be applied to previously wounded test areas and the surrounding skin (approx. 3 cm2). After a certain time the second skin biopsy will be taken from the treated test areas. The skin biopsies will be analysed via micro array.
  Arms: Arm 2

SUMMARY:
In previous in vitro studies it could be shown, that Dexpanthenol has an influence on the gene expression of fibroblasts. The genes which are influenced by Dexpanthenol play mainly a role during cell proliferating processes.The aim of this study is to investigate the molecular effect of Dexpanthenol on human living skin, during wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Skin type I to IV
* Willingness to avoid intensive sunlight exposure two weeks before the start of the study and at least 2 months after removal of the stitches

Exclusion Criteria:

* Active skin disease, moles, tattoos, strong pigmentation at the test area or scars in the test area that would influence the visual scoring
* History of keloids and hypertrophic scars
* Frequent visits of tanning booths
* Intake of drugs interfering with the immune system (e.g. antiphlogistics, corticosteroids, immunosuppressants, and antihistamines) within 30 days before day 1 as well as during the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2009-02; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Investigation of gene expression in dermal fibroblasts and keratinocytes on a molecular level. | Analysis of skin biopsies taken 24h, 72h and 144h after wounding

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Hamburg, Hamburg, Germany

REFERENCES:
- See also: Click here and search Bayer product information provided by the EMA — http://www.clinicaltrialsregister.eu